CLINICAL TRIAL: NCT06155695
Title: Targeting the Auditory Control Network With Auditory Control Enhancement (ACE) in Schizophrenia
Brief Title: Auditory Control Enhancement (ACE) in Schizophrenia
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian A Coffman, PhD (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Brian A Coffman, PhD, Research Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22070009; R21MH128823 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-12-04 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Auditory Hallucinations
MeSH Terms: conditions — Hallucinations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Auditory Control Enhancement (ACE) (Experimental): tDCS + ACCT
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Auditory Cognitive Control Training (ACCT)
- Sham tDCS + ACCT (Sham Comparator): Sham tDCS + ACCT
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Auditory Cognitive Control Training (ACCT)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS will be administered using the Starstim system. We will use the freely available Simulation of Non-Invasive Brain Stimulation (SimNIBS) software to optimally target the rVLPFC and left TPJ in each subject. Finite element models will be generated using T1 and T2 scans. We will generate multiple models to maximize on-target stimulation and minimize off-target stimulation, as determined by ratio of the summed current density within and beyond target regions of interest (ROIs). tDCS current in the active stimulation condition will be maintained at 2.0 milliamps (mA) for the first 45 minutes of each one-hour training session. Sham stimulation the same current, only the current will be ramped down to 0 mA after 30 seconds. Our previous research has shown this method to produce indistinguishable skin sensation. During tDCS, patients will be monitored for possible negative side effects.
Behavioral: Auditory Cognitive Control Training (ACCT) — ACCT incorporates a subset of components from Cognitive Enhancement Therapy found to have early benefits on the cognitive deficits of interest to the proposed studies and can be conducted more time-efficiently to achieve our specific goals. ACCT involves approximately 3 hours of computerized neurocognitive training using cognitive control and processing speed training software developed by Ben-Yishay and colleagues. Deficits in cognitive control are addressed with computer training exercises containing simple stimuli with little inherent emotional or motivational salience. ACCT requires individuals to be vigilant, inhibit irrelevant stimuli, and shift attention between auditory and visual modalities. Computer training exercises facilitate reaction time in a temporal mode using auditory cues (The Attention Reaction Conditioner), spatial focusing with visual cues (the Zero Accuracy Conditioner), and temporal vigilance with auditory and visual cues (Time Estimates).

SUMMARY:
The purpose of this clinical trial is to investigate neural markers of target engagement to further develop auditory control enhancement (ACE) as a novel, inexpensive, and noninvasive intervention to address treatment-refractory auditory hallucinations. Here, we will address questions about the feasibility and acceptability of ACE, as well as the degree to which ACE results in measurable engagement of biophysical and neurophysiological targets.

Participants will complete:

* Auditory Control Enhancement (ACE): Participants will be assigned by chance (such as a coin flip) into one of two groups to receive a different dosage or level of transcranial direct current stimulation (tDCS) during three sessions of cognitive training. tDCS is used to stimulate the brain for a short period of time. For tDCS one or two thin wet sponges are placed on the head and/or upper arm. The sponges will be connected to electrodes which will deliver a very weak electrical current. The Neuroelectrics Starstim 32 will be used to deliver tDCS.
* Interviews: Before and after ACE, in two separate sessions, participants will be asked questions about a) background; b) functioning in daily life and across different phases of your life and past, present and future medical records.
* Cognitive Tests: During the interview sessions, participants will also perform cognitive tests. Participants will be asked to complete computerized and pen-and-paper tests of attention, concentration, reading, and problem-solving ability.
* EEG scan: Participants will be asked to complete EEG (electroencephalography) studies before and after ACE training. EEG will be measured using the same Neuroelectrics Starstim 32 system used for tDCS. EEG measures the natural activity of the brain using small sensors placed on the scalp. These sensors use conductive gel to provide a connection suitable for recording brain activity. During EEG, participants will watch a silent video while sounds are played over headphones, or sometimes count the sounds. In addition to these auditory tasks, participants will also be asked to perform visual attention tasks, such pressing a button for a letter or image.
* Magnetic Resonance Imaging (MRI) Scan: Participants will also be asked to complete MRI studies before and after ACE training. An MRI is a type of brain scan that takes pictures of the brain that will later be used to create a 3D model of the brain. The MRI does not use radiation, but rather radio waves, a large magnet and a computer to create the images.

Researchers will compare individuals receiving ACE to those receiving sham tDCS during cognitive training to determine effects of ACE.

DETAILED DESCRIPTION:
Auditory hallucinations associated with schizophrenia (Sz) are pervasive, debilitating, and disturbing. Unfortunately, they are also difficult to treat - auditory hallucinations persist in about 25% of cases despite pharmacotherapy and treatment of cognitive symptoms (the symptoms most strongly related to global functioning) is modest at best. We propose a novel, inexpensive, and noninvasive intervention to address treatment-refractory symptoms, a critical need in Sz. Auditory hallucinations and impaired cognition in schizophrenia are not independent. Both are associated with system-level dysfunction of the fronto-temporal auditory control network, comprising auditory/verbal perceptual areas in temporoparietal junction (TPJ) and cognitive/behavioral control systems in ventrolateral prefrontal cortex (VLPFC). VLPFC traditionally inhibits and reattributes perceptual misrepresentations in most people. For those with schizophrenia, impairment of auditory cognitive control makes this impossible. Data from our lab suggest that auditory control network dysfunction may be central to the early etiology of the disorder. Auditory control enhancement (ACE) is designed to improve auditory control network function, thereby increasing inhibition of spurious auditory system activity in temporoparietal cortex and reducing auditory hallucinations. ACE combines a time-tested psychotherapeutic behavioral training program with targeted non-invasive brain stimulation using transcranial Direct Current Stimulation (tDCS). Our pilot data demonstrate the effectiveness of the behavioral training program and synergistic effects with tDCS of the auditory control network for treating treatment-refractory auditory hallucinations in schizophrenia. To further develop ACE for efficacy trials, we plan to investigate neural markers of target engagement in two sham-controlled experiments. Aim 1 will determine whether tDCS of right vlPFC (anode) and left TPJ (cathode) during MRI alters electric field measures and blood oxygenation level dependent (BOLD) response during stimulation to demonstrate that markers of tDCS current flow and BOLD fluctuate with induced current, and these fluctuations align spatially with computer models. Aim 2 will examine feasibility of subject retention and blinding for ACE. Aim 3 will examine the degree to which ACE modifies behavioral, neurophysiological, and hemodynamic markers of target engagement using neural oscillatory and cerebral blood flow (CBF) measures. Pilot data show feasibility of our aims and provide preliminary evidence that ACE has strong and lasting effects on auditory hallucinations assessed with the psychotic symptoms rating scale (PSYRATS), and that changes in cognitive factors associated with auditory hallucinations strongly correlate with changes in neural oscillatory measures of cognitive control. ACE represents a novel, transformative intervention with long-lasting effects that has the potential to change the treatment of schizophrenia and vastly improve the outcome for afflicted individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-40
* Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder, Psychosis not otherwise specified (NOS), Affective Psychosis with mood incongruent hallucinations.
* ability to provide informed consent
* Intelligence quotient (IQ) >= 70, as measured by the Weschler Abbreviated Scale of Intelligence (WASI)
* <5 years since the onset of first psychotic episode
* persistent auditory hallucinations without remission despite attempting >2 antipsychotic medications and having > 1 month of medication compliance

Exclusion Criteria:

* hearing deficit as assessed by audiometry (hearing threshold > 30 decibels (dB) nHL)
* standard MRI contraindications (e.g. cardiac pacemaker, aneurysm clip, cochlear implants, history of metal fragments in body, neurostimulators, weight of 300 lbs. or more, or claustrophobia)
* [self report] head injury with loss of conscious > 10 min, medical illness affecting brain function or structure, significant neurologic disorder (e.g. seizure disorder),
* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) substance use disorder - other than cannabis - and except individuals who have met at least early remission criteria (3 months without dependence symptoms) or a psychotic illness with a temporal relation to a substance use disorder
* currently pregnant or early postpartum (<6 weeks after delivery or miscarriage)
* currently taking medications that affect alertness, other than antipsychotic medication (e.g. sedatives, tranquilizers, muscle relaxants, and sleeping aids)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Magnetic field modulation with tDCS current | Week 1
  We will use General Linear Model (GLM) in SPM12 to assess the parametric modulation of 2nd-echo phase data with the applied tDCS current as a regressor. Magnetic field modulation of target areas will be quantified as the ratio of mean beta values within target areas in rVLPFC and left TPJ over the mean beta value over cortical voxels beyond these regions of interest.
Blood-Oxygen Level Dependent (BOLD) response modulation with tDCS current | Week 1
  We will use General Linear Model (GLM) in Statistical Parametric Modeling (SPM12) to assess the parametric modulation of 2nd-echo magnitude data with the applied tDCS current as a regressor. BOLD modulation within target areas will be quantified as the ratio of mean beta values within target areas in right ventrolateral prefrontal cortex (rVLPFC) and left temporoparietal junction (TPJ) over the mean beta value over cortical voxels beyond these regions of interest.
Change from baseline in oscillatory measure of cognitive control during stimulus evaluation in AX-CPT | Week 3 minus Week 1
  Mean event-related spectral power will be calculated between 300-500 ms after "A" and "B" stimuli in the gamma band (30-60 Hz), across frontocentral EEG electrodes (Fz, FC1, FCz, FC2). Cognitive control during stimulus evaluation will be quantified as the mean over "A" and "B" responses.
Change in oscillatory measure of cognitive control during response preparation in A-X version of the continuous performance test (AX-CPT) | Week 3 minus Week 1
  Mean event-related spectral power will be calculated between 600-1200 ms after "A" and "B" stimuli in the gamma band (30-60 Hz), across frontocentral EEG electrodes. Cognitive control during response preparation will be quantified as the difference between "A" and "B" responses (B minus A)).
Change in Auditory Steady-State Response (ASSR) Modulation with Attention | Week 3 minus Week 1
  Mean evoked event-related spectral power will be calculated between 100-500 ms after stimulus onset and 35-45 Hz in frontocentral electrodes (Fz, FC1, FCz, FC2). Attention modulation will be quantified as the difference between signal power measures in attend and ignore conditions (attend minus ignore).
Change in Auditory Steady-State Response (ASSR) amplitude. | Week 3 minus Week 1
  Mean evoked event-related spectral power will be calculated between 100-500 ms after stimulus onset and 35-45 Hz in frontocentral electrodes (Fz, FC1, FCz, FC2), from data recorded while participants ignore auditory stimuli.
Change in cerebral blood flow in auditory control regions | Week 3 minus Week 1
  Cerebral blood flow (CBF) measured by pseudo-continuous arterial spin labeling (pcASL) will be assessed in right vlPFC and left TPJ target regions
Retention | Through study completion, an average of 3 weeks
  Percentage of enrolled participants who did not complete the study
Blinding | Week 3
  Subjective forced-choice impression of treatment condition assessed by a single item on study completion questionnaire - "Which treatment condition do you think you received? ACE or sham(placebo)?"
Acceptability | Week 3
  Acceptability rating on a visual analogue scale (0-100; greater = more acceptable) obtained via post-study survey.

SECONDARY OUTCOMES:
Change in MCCB Attention Scale Score | Week 3 minus Week 1
  t-score (mean = 50, standard deviation= 10; greater=better) obtained on the Attention scale of the National Institute of Mental Health's Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS)- Consensus Cognitive Battery (MCCB)
Change in MCCB Processing Speed Scale Score | Week 3 minus Week 1
  t-score (mean = 50, SD = 10; greater=better) obtained on the Processing Speed scale of the MATRICS Consensus Cognitive Battery (MCCB)

OTHER OUTCOMES:
Change in Auditory Hallucination Severity | Week 3 minus Week 1
  Severity will be assessed using the PSYRATS (Physical scale; range = 0-4; greater = more severe)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Coffman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) collected in the trial, following deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication, and for at least 5 years
Access Criteria: Researchers who have access to NIH data archive will be able to access the data
URL: https://reporter.nih.gov/project-details/10593386

DOCUMENTS (1):
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT06155695/ICF_000.pdf